CLINICAL TRIAL: NCT07354646
Title: The Landscape of T1 Mapping for Disease Profiling in a Real-World Cohort
Brief Title: The Application of T1 Mapping in Real-World
Status: Recruiting | Type: Observational
Sponsor: Chinese Academy of Medical Sciences, Fuwai Hospital (Other)
Responsible Party: Principal Investigator, Minjie Lu, Department Director, Chinese Academy of Medical Sciences, Fuwai Hospital
Other Study IDs: CMR_T1 mapping
Record Dates: First submitted 2025-12-29; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Myocardial Infarction (MI); Hypertrophic Cardiomyopathy (HCM); Dilated Cardiomyopathy (DCM); Arrhythmogenic Cardiomyopathy; Myocarditis
MeSH Terms: conditions — Myocardial Infarction; Cardiomyopathy, Hypertrophic; Cardiomyopathy, Dilated; Myocarditis | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Healthy Controls: CMR criteria:
  Anatomically intact cardiac structures: LVEF, ventricular volumes, and wall thickness within sex- and BSA-adjusted reference ranges (LVEF ≥55%, LVEDVi <82 mL/m² for females, <97 mL/m² for males); Absence of pathological tissue characteristics (negative LGE); Normal hemodynamic profile: Competent valvular function without hemodynamically significant regurgitation or stenosis.
  Clinical exclusion criteria: No history of coronary artery disease, inflammatory cardiomyopathy, or electrophysiological abnormalities requiring intervention
  Interventions: Diagnostic Test: Magnetic Resonance Imaging with Contrast
- Myocardial Diseases: Patients with various myocardial diseases including Fabry disease, Iron-overload, atrial fibrillation (AF), hypertension, aortic stenosis (AS), chronic myocardial infarction (MI), acute MI, hypertrophic cardiomyopathy (HCM), dilated cardiomyopathy (DCM), restrictive cardiomyopathy (RCM), arrhythmogenic cardiomyopathy (ACM), acute myocarditis, chronic myocarditis, cardiac amyloidosis, cardiac tumor, congenital heart disease, and suspected transplant rejection.
  Interventions: Diagnostic Test: Magnetic Resonance Imaging with Contrast

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Imaging with Contrast — Participants in this arm undergo a single, standardized cardiac MRI scan with gadolinium-based contrast agent.

SUMMARY:
The goal of this observational study is to create a comprehensive real-world spectrum of T1 mapping measurements across different heart conditions. We aim to establish reference values for how heart tissue characteristics vary in various diseases, which will help doctors better interpret these advanced MRI measurements in clinical practice. The main questions it aims to answer are:

What are the normal T1 mapping values for different heart diseases, and how do they compare to healthy hearts? Can we use the simpler "native T1" measurement (without contrast dye) instead of the more complex "ECV" measurement (which requires contrast dye) for diagnosis?

Patients with various myocardial conditions will undergo CMR T1 mapping scans. We will analyze the MRI images and clinical records to establish disease-specific reference ranges for T1 mapping parameters, and validate the diagnostic accuracy of T1 mapping

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (≥18 years) with clinically diagnosed myocardial diseases based on current international guidelines.
2. Specific disease categories include:

   * Cardiomyopathies (HCM, DCM, RCM, ACM)
   * Infiltrative disorders (cardiac amyloidosis, Fabry disease)
   * Inflammatory conditions (acute/chronic myocarditis)
   * Ischemic heart disease (acute/chronic MI)
   * Valvular heart disease (aortic stenosis)
   * Arrhythmic conditions (atrial fibrillation)
   * Metabolic disorders (iron-overload)
   * Neoplastic conditions (cardiac tumors)
   * Congenital heart disease
   * Post-transplant evaluation
3. All diagnoses must be confirmed using established guideline-based criteria:

   * Echocardiographic parameters meeting disease-specific cutoffs
   * Cardiac MRI findings consistent with current consensus criteria
   * Laboratory biomarkers supporting respective diagnoses
   * Histopathological confirmation when clinically indicated

Exclusion Criteria:

* Presence of multiple cardiomyopathy diseases or risk factors simultaneously
* Contraindications to CMR examination
* Poor image quality precluding accurate T1 mapping analysis
* Incomplete clinical data for definitive diagnosis confirmation
* Pregnancy or lactation
* Inability to provide informed consent

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study population comprises a diverse cohort of patients with a comprehensive spectrum of myocardial conditions, including Fabry disease, iron overload, atrial fibrillation, hypertension, aortic stenosis, chronic and acute myocardial infarction, hypertrophic, dilated, restrictive, and arrhythmogenic cardiomyopathies, acute and chronic myocarditis, cardiac amyloidosis, cardiac tumors, congenital heart disease, and cases of suspected transplant rejection. This population represents a wide array of pathophysiological processes affecting the myocardium, ensuring broad clinical relevance and generalizability of the study findings.
Sampling Method: Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-03-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Ranges of T1 mapping values | From enrollment until completion of the last T1 mapping examination, assessed up to 5 years

CONTACTS AND LOCATIONS:
Locations (1):
- Fuwai Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No